CLINICAL TRIAL: NCT02681237
Title: A Proof of Concept, Multi-centre, Clinical Trial of the Combination Cediranib-Olaparib at the Time of Disease Progression on PARP Inhibitor in Ovarian Cancer
Brief Title: A Study of Cediranib and Olaparib at Disease Worsening in Ovarian Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: e-Volve 1
Record Dates: First submitted 2016-02-10; First posted 2016-02-12 (Estimated); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — cediranib; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cediranib and Olaparib (Experimental): Cediranib will be given by mouth, at a dose of 20 mg, once a day, everyday.
  Olaparib will given by mouth, at a dose of 300 mg, twice a day, every day.
  Interventions: Drug: Cediranib; Drug: Olaparib

INTERVENTIONS:
Drug: Cediranib — Small-molecule inhibitor of several tyrosine kinases including VEGFR-1, VEGFR-2, VEGFR-3 and c-kit.
Drug: Olaparib — Poly (ADP-ribose) polymerase (PARP) inhibitor.

SUMMARY:
This is a proof of concept study (a study to initially assess the benefit a new drug indication) of the combination of two investigational drugs cediranib and olaparib in patients with ovarian cancer whose cancer worsened despite previously receiving a poly (ADP-ribose) polymerase (PARP) inhibitor (such as olaparib).

The purpose of this study is to find out whether taking cediranib and olaparib at the same time will be able to stop tumors from growing further or shrink it.

Cediranib works by blocking (inhibiting) several specific proteins in cancer cells called the vascular endothelial growth factor (VEGF) receptors. These proteins are important in the formation of blood vessels to the tumor. It is believed that many tumors survive because the blood vessels on the tumors bring oxygen and nutrients to the cancer cells which enable them to grow. If the formation of the blood vessels is blocked, the tumor cells may die.

Olaparib, works by blocking a protein called poly [adenosine diphosphate-ribose] polymerase (PARP). PARP is an important protein which tries to fix damaged deoxyribonucleic acid (DNA, molecules that contain important instructions for the development of cells). Many cancers are thought to develop from damaged DNA. By blocking PARP from fixing damaged DNA, the tumor cells may die.

Adding cediranib to olaparib, and therefore blocking several different mechanisms for cancer growth, may stop tumor growth.

DETAILED DESCRIPTION:
The recent changes in OC treatment with maintenance therapy raise the question of drug strategy at progression. It remains unclear what the best option for a patient relapsing during PARP inhibitor treatment would be. Findings from a retrospective study-and the first data available for treatment after a PARP inhibitor-have provided support for a lack of significant clinical cross-resistance between PARP inhibitor and platinum-based chemotherapy. However, based on a recent clinical trial, the addition of an anti-angiogenic to olaparib adds significant benefit. In a randomized phase II trial, cediranib with olaparib showed an objective response rate markedly higher in the combination arm (80%) than the olaparib single agent arm (48%) with a median PFS of 9.0 months for olaparib and 17.7 months for cediranib/olaparib (p=0.001). The overall rate of grade 3/4 toxicity was higher on the combination (70%) than on olaparib (7%). The main toxicities occurring were fatigue (27% cediranib/olaparib vs 7% olaparib), diarrhea (23% vs 0%), and hypertension (39% vs 0%). This is the first oral, non-chemotherapy-based combination treatment in the platinum-sensitive recurrent OC. Preclinically, PARP-inhibition has reported anti-angiogenic effects, where GPI 15427 (a potent PARP-1/2 inhibitor) inhibits in vivo angiogenesis in a matrigel plug assay. PARP-1 knockout mice also demonstrate decreased in vivo angiogenesis compared to control mice with wild-type PARP-1, supporting the notion that the observed anti-angiogenic effects are specific to anti-PARP activity. More recent work has demonstrated that HR can be suppressed by hypoxia through downregulation of HR repair proteins such as BRCA1 and RAD51 and that PARP inhibitor sensitivity is enhanced in hypoxic states. This information raises the hypothesis that PARP-inhibitors and anti-angiogenics may have synergistic effects. Furthermore, preclinical data demonstrated that hypoxia-mediated defects in DNA repair can lead to genetic instability and drive oncogenesis. Some patients with tumor expressing a 'mutator' phenotype due to the acquisition of repair-deficient cancer cells from an unfavourable tumour microenvironment could benefit from this combined approach. Based on evidence for targeting HRR and angiogenesis (two potential Achilles Heels in OC), we will evaluate the interest in adding cediranib to olaparib in patients relapsing after initial good response to olaparib treatment. This is a proof of concept study as we will assess the benefit of adding cediranib to olaparib at the time of disease progression under olaparib. As other PARP inhibitor are currently under investigations such as Rucaparib and ABT-888, with no data available regarding a rechallenge of PARP inhibitor beyond progression, we propose the combination cediranib and olaparib in the setting of disease progression under treatment with a PARP inhibitor such as olaparib.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years.
* Performance status <= 2.
* Histologically confirmed ovarian cancer, high grade serous or high grade endometrioid histology subtype.
* Radiographically documented disease progression within 28 days of registration and evaluable.
* Radiological progression on any PARP inhibitor therapy (example: olaparib):

  * a cohort of platinum sensitive recurrence and response for at least 6 months on PARP inhibitor treatment
  * a cohort of platinum resistance with disease progression within 6 months after the last dose of a platinum based chemotherapy
* Patients who discontinue PARP therapy will be eligible after a break in therapy or intervening therapy.
* Patients must have adequate bone marrow, renal and hepatic function per local laboratory reference range.
* Ongoing prior toxicities related to previous treatments must be recovered to <= grade 2 at the time of registration.
* Left ventricular ejection fraction (LVEF) >= 50% by echocardiograms or multigated acquisition (MUGA) scan within 28 days of registration.
* Acceptable urine dipstick/urine analysis for proteinuria.
* Patients are willing to undergo tumour biopsy pre-treatment if a biopsy at the time of progression on olaparib is not available.
* Life expectancy of greater than 3 months.
* Ability to understand and the willingness to sign a written informed consent document.
* Patient's willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
* Patients of child bearing potential and their partners who are sexually active must agree to the use of 2 highly effective forms of contraception throughout their participation during the study treatment and for 3 months after last dose of study treatment(s).

Exclusion Criteria:

* Patients with current bowel obstruction.
* Patients with known brain metastases.
* Unacceptable mean corrected QT (QTc) in screening electrocardiograms within 7 days of registration or history of familial long QT syndrome.
* Uncontrolled intercurrent illness including, but not limited to hypertension, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* A New York Heart Association classification of III or IV.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to olaparib or cediranib.
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Patients with myelodysplastic syndrome/acute myeloid leukaemia.
* Immuno-compromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV), patients with known active hepatitis (i.e., hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids.
* Patients who require maximal doses of calcium channel blockers to stabilize blood pressure.
* Patients with significant hemorrhage or haemoptysis.
* Patients who have had recent (within 2 weeks of registration, or until any wound has completely healed) major thoracic or abdominal surgery prior to study start, or a surgical incision that is not fully healed.
* History of stroke or transient ischemic attack within six months.
* Patients that are receiving and cannot stop the following prohibited medications prior to Cycle 1, Day 1.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-04-29 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | 8 weeks
  objective response rate by RECIST 1.1
Progression-Free Survival Rate | 16 weeks
  objective response rate by RECIST 1.1 or death

SECONDARY OUTCOMES:
CA125 response rate | 2 years
  objective response rate by GCIG criteria
Disease control rate | 2 years
Overall survival rate | 2 years
Number of Adverse Events Experienced | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Amit Oza, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lheureux S, Oaknin A, Garg S, Bruce JP, Madariaga A, Dhani NC, Bowering V, White J, Accardi S, Tan Q, Braunstein M, Karakasis K, Cirlan I, Pedersen S, Li T, Farinas-Madrid L, Lee YC, Liu ZA, Pugh TJ, Oza AM. EVOLVE: A Multicenter Open-Label Single-Arm Clinical and Translational Phase II Trial of Cediranib Plus Olaparib for Ovarian Cancer after PARP Inhibition Progression. Clin Cancer Res. 2020 Aug 15;26(16):4206-4215. doi: 10.1158/1078-0432.CCR-19-4121. Epub 2020 May 22. PMID 32444417